CLINICAL TRIAL: NCT03113682
Title: A Pilot Study of Cognitive-Behavioral Therapy for Rumination Disorder
Brief Title: A Study of Cognitive-Behavioral Therapy for Rumination Disorder
Acronym: CBT-RD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1702005190
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Rumination Disorder
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: There is only one arm in this study - all participants will be in the same arm, as all participants will receive CBT-RD. There is no control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (CBT-RD) (Experimental): There is only one arm in this study - all participants will be in the same arm, as all participants will receive CBT-RD. There is no control group.
  Interventions: Behavioral: CBT-RD

INTERVENTIONS:
Behavioral: CBT-RD — 5-8 sessions of cognitive behavioral therapy for rumination disorder (CBT-RD), held once per week in an outpatient setting.

SUMMARY:
The primary aim of this study is to pilot cognitive behavioral therapy (CBT-RD) for 10 individuals ages 10 and older who have rumination disorder

DETAILED DESCRIPTION:
Rumination disorder (RD; also known as "rumination syndrome") is a disordered eating behavior characterized by the repeated regurgitation of food during or soon after eating. The frequency of repeated regurgitation of food typically occurs at least a few times per week, frequently daily with subsequent re-chewing, re-swallowing, or spitting out of the regurgitated material. The widely used technique for treatment of RD has typically been diaphragmatic breathing, which works by serving as a competing response to abdominal wall contractions, which is hypothesized to trigger regurgitation. However, the efficacy of diaphragmatic breathing remains unknown and has mainly been delivered through a one-session instruction with an occasional follow-up.

In the absence of evidence-based treatments for RD, the investigators, alongside a collaboration with Dr. Jennifer Thomas at the Eating Disorders Clinical and Research Program (EDCRP) at Massachusetts General Hospital, have created a manualized treatment, Cognitive-Behavioral Therapy for Rumination Disorder (CBT-RD) informed by published case reports and currently in use at EDCRP at Massachusetts General Hospital and the Psychological Services Center at Drexel University. CBT-RD targets the habitual contraction of the abdominal wall and preceding events through the use of habit reversal, using primarily diaphragmatic breathing as a competing response.

This study involves a phone screen to determine eligibility, followed by 5-8 sessions of CBT-RD (approximately 50 minutes each). A battery of questionnaires will be administered at pre-treatment, post-treatment, and 3-month follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 or above
* Experience repeated regurgitation of food during or soon after eating, consistent with rumination disorder
* If applicable, have stable psychiatric medication for the past three months

Exclusion Criteria:

* Currently engage (in past three months) in any regular compensatory behaviors (e.g., self-induced vomiting, laxative/diuretic use)
* Current diagnosis of anorexia nervosa
* Acute suicide risk
* Are currently receiving psychological treatment for rumination disorder
* Co-morbid clinically significant psychological disorder that would require attention beyond the study treatment (e.g., psychotic disorder, substance dependence)
* Current pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Pica, Avoidant/Restrictive Food Intake Disorder, Rumination Disorder Interview (PARDI) | Change from baseline to 3-month follow-up
  A semi-structured interview to assess pica, Avoidant/Restrictive Food Intake Disorder (ARFID), and/or rumination disorder diagnosis, severity, and symptoms. We will use the PARDI to assess frequency and severity of rumination behavior specifically.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States